CLINICAL TRIAL: NCT00503529
Title: Open-label Phase IV Study to Investigate the Seropersistence of Tick Borne Encephalitis (TBE) Virus Antibodies After the First Booster and the Response to a Second Booster Vaccination With FSME-IMMUN 0.5ml in Adults (Follow Up to Study 223)
Brief Title: TBE Antibody Persistence and Booster Vaccination Study in Adults (Follow-up to Study 223)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 690701; EUDRACT # 2007-000440-27
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Encephalitis, Tick-Borne
MeSH Terms: conditions — Encephalitis, Tick-Borne | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Tick-Borne Encephalitis (TBE) Vaccine (Inactivated) — Vaccination by intramuscular injection into the right or left upper arm (musculus deltoideus)
  Other Names: FSME-IMMUN 0.5 ml

SUMMARY:
The purpose of this study is to assess:

* TBE antibody persistence 24, 34, 46 and 58 months (as applicable) after the first booster TBE vaccination with FSME-IMMUN 0.5ml given in Study 223, by means of ELISA (IMMUNOZYM FSME IgG) and Neutralization test (NT),
* TBE antibody response to a second booster vaccination with FSME-IMMUN 0.5ml in the present study, by means of ELISA and NT,
* Safety of FSME-IMMUN 0.5ml after the second booster vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who participated in Study 223 will be eligible for participation in this study if:
* they understand the nature of the study, agree to its provisions and provide written informed consent
* they received the first booster vaccination with FSME-IMMUN 0.5ml during the course of study 223
* blood was drawn after their first booster vaccination in Study 223.

Exclusion Criteria:

Subjects will be excluded from participation in this study if they:

* received any TBE vaccination since their first booster vaccination with FSME-IMMUN 0.5ml
* have a history of infection with or vaccination against other flaviviruses (e.g. dengue fever, yellow fever, Japanese B-encephalitis) since their first booster vaccination with FSME-IMMUN 0.5ml
* are known to be HIV positive (a special HIV test is not required for the purpose of the study) since their first booster vaccination with FSME-IMMUN 0.5ml
* have a known or suspected problem with drug or alcohol abuse (> 4 liters wine / week or equivalent level of other alcoholic beverages).

Subjects will not be eligible for booster vaccination if they:

* are not clinically healthy, (i. e. the physician would have reservations vaccinating with FSME-IMMUN 0.5ml outside the scope of a clinical trial)
* suffer from a disease (e.g. autoimmune disease) or are undergoing a form of treatment (e.g. systemic corticosteroids) that can be expected to influence immunological functions
* are females of childbearing potential and are pregnant or breastfeeding before the booster vaccination (positive pregnancy test result at the medical examination before the booster vaccination)
* have shown an allergic reaction to one of the components of the vaccine since their first booster vaccination in Study 223
* are simultaneously participating in another clinical trial including administration of an investigational product within six weeks prior to the booster vaccination until the end of the study
* do not agree to keep a Subject Diary.
* Subjects who meet the eligibility criteria, but have a febrile illness (body temperature >= 38.0°C, measured orally) at the scheduled time of vaccination, will not be vaccinated until their body temperature returns to normal.
* Subjects who have been administered any vaccination within 2 weeks prior to the booster vaccination will not be vaccinated until an interval of two weeks has passed.
* If subjects have received antipyretics within 4 hours prior to the scheduled time of vaccination, the vaccination should be performed at a later time.
* If a subject had a tick-bite within 4 weeks of the scheduled booster vaccination, the vaccination shall be delayed such that an interval of 4 weeks has passed since the tick-bite in order to avoid any interference with diagnostic assays in the event of a TBE infection.
* If a subject has donated blood or plasma or has received a blood transfusion or immunoglobulins within 4 weeks of the scheduled booster vaccination, the vaccination shall be delayed until an interval of 4 weeks has passed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2007-07; Primary Completion 2010-07 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Seropositivity rate measured by Enzyme-Linked Immunosorbent Assay (ELISA) and/or Neutralization test (NT) 24, 34, 46 and 58 months after the first booster TBE vaccination in Study 223 and after the booster vaccination in this study | 24, 34, 46 and 58 months after the the first booster TBE vaccination in Study 223 and after the booster vaccination in this study (study ID 690701)

CONTACTS AND LOCATIONS:
Overall Officials: Ryszard Konior, MD, Principal Investigator — The John Paul II Hospital, Krakow, Poland
Locations (2):
- Poland (2):
  - Hospital in Debica - Zespol Opieki Zdrowotnej w Debicy, Dębica
  - Szpital Jana Pawla II (The John Paul II Hospital) Oddzial Neuroinfekcji, Krakow

REFERENCES:
- [Derived] Konior R, Brzostek J, Poellabauer EM, Jiang Q, Harper L, Erber W. Seropersistence of TBE virus antibodies 10 years after first booster vaccination and response to a second booster vaccination with FSME-IMMUN 0.5mL in adults. Vaccine. 2017 Jun 16;35(28):3607-3613. doi: 10.1016/j.vaccine.2017.03.059. Epub 2017 May 22. PMID 28545923